CLINICAL TRIAL: NCT05717673
Title: Effect of Epi-Off Technique in Corneal Collagen Cross Linking On Endothelial Count by Using Specular Microscopy in Keratoconus Patients
Brief Title: Effect of Epi-Off Technique Corneal CXL On Endothelial Count by Specular Microscopy in Keratoconus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heba Allah Nashaat Mohamed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Heba Allah Nashaat Mohamed, Determine safety of CXL on corneal endothelial count by using specular microscopy in patients with keratoconus, Assiut University
Organization: Assiut University (Other)
Other Study IDs: EOEOCXLOEnCBsMK
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Keratoconus, Collagen
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Specular microscopy — Specular microscopy is a noninvasive photographic technique that analyze the corneal endothelium. Using computer-assisted morphometry, modern specular microscopes analyze the size, shape and population of the endothelial cells. The instrument projects light onto the cornea and captures the image that is reflected from the optical interface between the corneal endothelium and the aqueous humor. The reflected image is analyzed by the instrument and displayed as a specular photomicrograph

SUMMARY:
Determine safety of EPi-off CXL on corneal endothelium by using specular specular microscopy to assess endothelial count.

DETAILED DESCRIPTION:
Specular microscopy is a noninvasive photographic technique that analyze the corneal endothelium. Using computer-assisted morphometry, modern specular microscopes analyze the size, shape and population of the endothelial cells. The instrument projects light onto the cornea and captures the image that is reflected from the optical interface between the corneal endothelium and the aqueous humor. The reflected image is analyzed by the instrument and displayed as a specular photomicrograph

Corneal collagen cross-linking (CXL) is a therapeutic procedure aiming at increasing the corneal stiffness in the keratoconus eyes by induction of cross-links within the extracellular matrix. It is achieved by ultraviolet-A (370 nm) irradiation of the cornea after saturation with the photosensitizer riboflavin. In the conventional CXL protocol, a minimum (manual) de-epithelialized corneal thickness of 400 μm is recommended to avoid potential irradiation damage to the corneal endothelium. In advanced keratoconus, however, stromal thickness is often lower than 400 μm, which limits the application of CXL in that category. Efforts have been undertaken to modify the conventional CXL procedure to be applicable in thin corneas. The current review discusses different techniques employed to achieve this end and their results. The overall safety and efficacy of the modified CXL protocols are good, as most of them managed to halt the progression of keratectasia without postoperative complications. However, the evidence of safety and efficacy in the use of modified CXL protocols is still limited to few studies with few patients involved. Controlled studies with long-term follow-up are required to confirm the safety and efficacy of it.

ELIGIBILITY:
Inclusion Criteria:

* Patients with corneal diseases that treated by collagen cross linking such as keratokonus and post lasic ectesia with corneal thickness above 400um at its thinnest location.

Exclusion Criteria:

1. Prior herpetic infection
2. Autoimmune disorders
3. corneal thickness below 400um at its thinnest location
4. Corneal opacity

Ages: 10 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People have keratoconus from 10 years to 75 years has corneal thickness more than 400 um at the thinnest location of the cornea with exclusion criteria like prior herpetic infection or autoimmune disease or corneal opacity
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-05 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Determine safety of CXL on corneal endothelial count by using specular microscopy in patients with keratoconus | 6 months
  by using specular microscopy to assess endothelial count to prevent corneal damages

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aly Momen, Study Director — Assiut University
Locations (1):
- Assuit university, Asyut, Egypt